CLINICAL TRIAL: NCT04797195
Title: Improving Care for Peritoneal Dialysis Patients With the CKD-PD App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Khon Kaen University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Katharine E. Morley, Associate Physician, Department of Medicine, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018A013145; 1R21TW010963-01A1 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Kidney Failure, Chronic; Peritoneal Dialysis Complication
Keywords: mobile health; peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-PD app user group (Experimental): Patients on peritoneal dialysis using the CKD-PD app and home monitoring equipment to measure and record blood pressure, body weight, and dialysis fluid removed
  Interventions: Other: CKD-PD app with home monitoring equipment
- Usual care group (No Intervention): Patients on peritoneal dialysis using handwritten notebook to record record blood pressure, body weight, and dialysis fluid removed; measurements obtained through usual method

INTERVENTIONS:
Other: CKD-PD app with home monitoring equipment — use home monitoring equipment to measure blood pressure, body weight, and dialysate fluid volume and record in CKD-PD app
  Arms: CKD-PD app user group

SUMMARY:
Managing the hydration status in patients undergoing peritoneal dialysis (PD) is a key task for nephrologists in Thailand that is made difficult due to lack of timely access to hydration metrics including weight, blood pressure, and ultrafiltration volume. This research project aims to improve the monitoring of hydration status in PD patients from a bimonthly, in-clinic review of a handwritten log-book to a smart phone based app (CKD-PD) with digitized data that allows for near real time monitoring hydration abnormalities, thereby creating the opportunity for earlier treatment of overhydration. The investigators hypothesize that use of the CKD-PD will improve early treatment of overhydration, and potentially reduce the incidence of complications, hospitalizations, and mortality in PD patients.

DETAILED DESCRIPTION:
The number of patients in Thailand with end stage renal disease on peritoneal dialysis (PD) is growing rapidly. Thai nephrologists have identified a critical gap in the current management of PD patients: a lack of timely information about fluid (hydration) status. Real time access to this information creates the opportunity for the early treatment of overhydration - the most common cause of complications and hospitalization in this population. Early treatment of overhydration in PD patients can decrease the incidence of complications, improve quality of life, and decrease health care costs.

This research project aims to improve the monitoring of fluid status in PD patients from a bimonthly, in-clinic review of handwritten log books to a smart phone based app ("CKD-PD") with digitized data. This allows for near real time data visualization, hydration status monitoring, outlier notifications, and more timely treatment interventions for overhydration. Data from home monitoring equipment to transferred to the CKD-PD app. Hydration metrics are uploaded to "CKDNET" (Chronic Kidney Disease NorthEast Thailand) database in the Thai Care Cloud - Thailand's national health database, merging patient collected data with hospital and clinic records.

The objective of this study is to determine if use of the CKD-PD app can improve early treatment of overhydration in PD patients. The investigators will conduct a randomized clinical trial comparing the incidence of clinical interventions for treatment of overhydration. PD patients from 3 facilities in Northeast Thailand - Srinagarind Hospital at Khon Kaen University, Khon Kaen Hospital and Chaiyaphum Hospital - (N=200) will be randomized into two groups - one using the CKD-PD app, and one receiving usual management. The primary outcome will be the incidence of clinical intervention to treat overhydration as an intermediate outcome related to the secondary outcomes: complications, hospitalizations, and mortality related to fluid overload.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease from any cause on home based peritoneal dialysis
* age greater than 18 years
* access to a smart phone capable of running the CKD-PD app

Exclusion Criteria:

* vulnerable populations including children, prisoners, pregnant women, individuals with cognitive impairment, refugees
* unwillingness to sign consent or participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine E Morley, MD, MPH, Principal Investigator — Massachusetts General Hospital; Sirirat Anutrakulchai, MD PhD, Principal Investigator — Srinagarind Hospital, Khon Kaen University
Locations (3):
- Thailand (3):
  - Chaiyaphum Hospital, Chaiyaphum
  - Khon Kaen Hospital, Khon Kaen
  - Srinagarind Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anutrakulchai S, Tatiyanupanwong S, Kananuraks S, Lukkanalikitkul E, Kongpetch S, Chotmongkol W, Morley MG, Thinkhamrop W, Thinkhamrop B, Kleebchaiyaphum C, Khianchanach K, Chunghom T, Morley KE. Effect of the Chronic Kidney Disease-Peritoneal Dialysis (CKD-PD) App on Improvement of Overhydration Treatment in Patients on Peritoneal Dialysis: Randomized Controlled Trial. J Med Internet Res. 2025 May 21;27:e70641. doi: 10.2196/70641. PMID 40397925

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CKD-PD App User Group | Usual Care Group
Started | 103 | 105
Completed | 77 | 73
Not Completed | 26 | 32
Not completed — Death | 8 | 15
Not completed — Change from PD | 15 | 15
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CKD-PD App User Group | Usual Care Group | Total
Number analyzed (Participants) | 103 | 105 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (15.5) | 54.8 (14.8) | 54.3 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 54 | 117
  Male | 40 | 51 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 103 | 105 | 208
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 103 | 105 | 208
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 103 | 105 | 208
Hospital [Count of Participants; unit: Participants]
  Srinagarind | 20 | 20 | 40
  Khon Kaen | 35 | 37 | 72
  Chaiyaphum | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Clinical Interventions for Over Hydration
Description: Change in treatment in response to over hydration detected by clinical symptoms or abnormal hydration metrics. Includes change in antihypertensive or diuretic medications, change in dialysis prescription, fluid/salt dietary change, referral to clinic for evaluation or hospitalization
Time Frame: through study completion, average 1 year
Measure: Number; unit: clinical interventions
Arm/Group | CKD-PD App User Group | Usual Care Group
Number analyzed (Participants) | 103 | 105
clinical interventions | 473 | 164

2. Secondary Outcome: Complication of Over Hydration Requiring Hospitalization
Description: Clinical event due to over hydration requiring hospitalization. Includes volume overload, infections, peritonitis, major adverse cardiac event, severe hypertension or stroke
Time Frame: through study completion, average 1 year
Measure: Number; unit: events
Arm/Group | CKD-PD App User Group | Usual Care Group
Number analyzed (Participants) | 103 | 105
events | 67 | 113

3. Secondary Outcome: Technique Failure
Description: Inability to continue peritoneal dialysis for any reason requiring a change to hemodialysis
Time Frame: through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CKD-PD App User Group | Usual Care Group
Number analyzed (Participants) | 103 | 105
Participants | 14 | 15

4. Secondary Outcome: Mortality
Description: Deaths occuring during study period for any cause
Time Frame: through study completion, average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CKD-PD App User Group | Usual Care Group
Number analyzed (Participants) | 103 | 105
Participants | 8 | 15

5. Other Pre Specified Outcome: Clinic Contacts
Description: Communication by phone or messaging app between peritoneal dialysis patients or surrogate regarding clinical concern about symptoms or hydration metrics
Time Frame: through study completion, average 1 year
Measure: Number; unit: events
Arm/Group | CKD-PD App User Group | Usual Care Group
Number analyzed (Participants) | 103 | 105
events | 473 | 164

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period for each individual, with a median follow up time in the app group of 11.2 months and non-app group of 11 months
Description: Adverse events were considered to be deaths, technique failure (change from peritoneal dialysis to another form of renal replacement therapy), and all cause hospitalizations.
  Patients undergoing peritoneal dialysis have frequent occurrences of death, technique failure and hospitalizations at baseline
Arm/Group | CKD-PD App User Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 8/103 | 15/105
Serious Adverse Events (participants affected / at risk) | 54/103 | 75/105
Other Adverse Events (participants affected / at risk) | 0/103 | 0/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CKD-PD App User Group (N=103) | Usual Care Group (N=105)
Technique failure (Renal and urinary disorders) | 14 (14) | 15 (15) — Unable to continue on peritoneal dialysis due to complications such as catheter malfunction, recurrent peritonitis, inadequate dialysis
Hospitalizations (General disorders) | 40 | 60 — All cause hospitalizations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT04797195/Prot_SAP_ICF_000.pdf